CLINICAL TRIAL: NCT06779539
Title: A Study of Ensartinib as Neoadjuvant Therapy for Patients With ALK Positive Resectable Stage II to III Non-Small Cell Lung Cancer：A Prospective, Open-label, Multi-center, Single-arm, Phase II Clinical Trial
Brief Title: Neoadjuvant Ensartinib in ALK Positive Resectable Stage II to III Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Zhou Qinghua, Professor of Surgical Oncology and Molecular Biology, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOG-0003
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ensartinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ensartinib (Experimental)
  Interventions: Drug: Ensartinib

INTERVENTIONS:
Drug: Ensartinib — Ensartinib 225 mg oral once daily 12 weeks

SUMMARY:
This single-arm, prospective, multicenter, phase II study is designed to evaluate the efficacy and safety of ensartinib as neoadjuvant treatment in ALK positive, resectable for stage II to III non-small cell lung cancer patients.

DETAILED DESCRIPTION:
This is a single-Arm, prospective, multicenter, phase II study, the primary endpoint is pathological complete response (pCR). Participants will receive ensartinib at 225 mg orally once a day taken with or without food for 12 weeks before surgical resection.

ELIGIBILITY:
Inclusion Criteria:

1. Give written informed consent before any study procedure.
2. Male or female aged between 18 and 75 years old (including 18 and 75 years old).
3. Histologically or cytologically documented lung adenocarcinoma within 60 days prior to study enrollment.
4. Clinical stage II-III assessed by EBUS-TBNA or PET/CT can be resected.
5. Patients confirmed as ALK fusion positive by RBK (NGS) test.
6. Presence of at least one accurately measurable lesion, CT showing a maximum diameter of 10mm at baseline (except for lymph nodes with a short axis of 15mm required) and suitable for accurate repeat measurements.
7. Eastern Cooperative Oncology Group (ECOG) performance status （PS） of 0 or 1.
8. Adequate hematological, biochemical and organ functions, defined as follows

   1. Hemoglobin ≥90g/L. Note: transfusions are allowed to meet the required hemoglobin level;
   2. Absolute neutrophil count (ANC) ≥1.5× 10^9/L
   3. Platelets ≥90 × 10^9/L;
   4. Total bilirubin ≤ 2 times the upper limit of normal (ULN)；
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5× ULN;
   6. Creatinine ≤ 1.5× ULN and creatinine clearance ≥ 60 mL/min.
9. Cardiopulmonary function suitable for surgical treatment (ECG, echocardiography, pulmonary function or blood gas analysis);
10. At least 2 weeks prior to initial trial treatment female subjects should use adequate contraceptive measures, the pregnancy test must be negative and there is no ongoing breastfeeding. Otherwise, one of the following criteria must be met during screening to prove the possibility of no fertility:

    1. Postmenopausal is defined as amenorrhea for at least 12 months after stopping all exogenous hormone treatment over 50 years old;
    2. Women under the age of 50 should be regarded as menopause if they stop menopause for 12 months or more after stopping exogenous sex hormone therapy, and their LH and FSH levels are within the postmenopausal range of the institution;
    3. Irreversible surgical sterilization recorded by hysterectomy, bilateral oophorectomy or bilateral salpingectomy, but excluding tubal ligation.
11. Men with partners of childbearing potential willing to use adequate contraceptive measures during the study and for 3 months after the last dose of study medication.

Exclusion Criteria:

1. Mixed squamous cell carcinoma, large cell neuroendocrine carcinoma or small cell lung cancer;
2. Prior treatment with any anti-cancer therapy;
3. Pregnant female patients; breastfeeding female patients.
4. Current use of (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4 (at least 3 weeks prior). All patients must try to avoid using or ingesting any drugs, herbal supplements and/or foods that are known to have induced effects on CYP3A4.
5. Evidence of any severe or uncontrolled systemic disease, including uncontrolled hypertension and active bleeding, that the investigator considers to be detrimental to patient participation in the study or to adherence to the protocol. Active and clinically significant bacterial, fungal, or viral infection including hepatitis B virus (HBV) or hepatitis C virus (HCV) or known human immunodeficiency virus (HIV). Screening for chronic diseases is not a requirement.
6. Past medical history of Interstitial lung disease（ILD）, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
7. A history of hypersensitivity to active or inactive excipients of Ensartinib or to drugs of similar chemical structure or class to Ensartinib, and uncontrollable nausea and vomiting, chronic gastrointestinal disease, inability to swallow drugs, or had undergone major bowel resection that would interfere with adequate absorption of Ensartinib.
8. Any of the following cardiac criteria:

   1. Mean resting corrected QT interval (QTc)>470 msec, obtained from 3 electrocardiograms (ECGs)
   2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG e.g., complete left bundle branch block, third-degree heart block, second-degree heart block.
   3. Any factors that increase the risk of QTc prolongation or the risk of arrhythmic events such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval.
9. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia；
10. Other circumstances deemed inappropriate by the investigator for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2028-06-12 (Estimated); Study Completion 2030-12-12 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | Within 2 month after surgery
  pCR rate is defined as the proportion of participants who have achieved pathologic complete response (with no residual viable tumor in lung primary or lymph nodes as evaluated by central pathology laboratory of surgical specimens) in all participants.

SECONDARY OUTCOMES:
Major Pathological Response (MPR) rate | Within 2 month after surgery
  MPR rate is defined as the proportion of participants who have achieved major pathologic response (less than or equal to 10% of residual viable tumor in lung primary or lymph nodes as evaluated by central pathology laboratory of surgical specimens) in all participants.
Objective Response Rate (ORR) | Pre-operation
  ORR was defined as the percentage of participants who attained complete response (CR) or partial response (PR). Responses are according to RECIST 1.1 as assessed by investigator.
Incidence of Adverse Events | Up to 1 month after surgery
  Toxicity will be graded by NCI Common Terminology Criteria for Adverse Events (CTCAE version 5.0)
Disease free survival (DFS) | 3 years postoperatively
  DFS is defined as the time from the first day after radical surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
Overall Survival (OS) | 5 years postoperatively
  OS was defined as the time from the date of enrollment to death from any cause.